CLINICAL TRIAL: NCT06437925
Title: Effects of the Use of Probiotics Ayran on Gingival Inflammation: An Experimental Gingivitis Study
Brief Title: Effects of Probiotic Ayran on Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cenk Haytac, Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Cukurova University-1
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Gingivitis; Probiotics; Inflamed Gums
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic ayran drink (Experimental): The participants in this experimental group will use probiotic containing ayran for 42 days and then will be subjected to 5 days of experimental gingivitis.
  Interventions: Dietary Supplement: probiotic ayran drink
- Placebo ayran drink (Placebo Comparator): The participants in this control group will use control ayran without probiotics for 42 days and then will be subjected to 5 days of experimental gingivitis.
  Interventions: Dietary Supplement: Placebo ayran drink

INTERVENTIONS:
Dietary Supplement: probiotic ayran drink — The test group has received probiotic ayran drink for 6 weeks
  Arms: Probiotic ayran drink
Dietary Supplement: Placebo ayran drink — The control group has received placebo ayran drink for 6 weeks
  Arms: Placebo ayran drink

SUMMARY:
Objectives: This study investigates the effects of daily consumption of probiotic ayran drink on gingival inflammation and the development of experimental gingivitis.

Methods: A total of 54volunteer students were included in the present randomized, double-blind, placebo-controlled trial.The participants were divided randomly into two groups; The Control group consisted of 27 participants who consumed placebo ayran, while the 27 participants of the Test group consumed probiotic ayran (containing Lactobacillus acidophilus and Bifidobacterium bifidum) for 42 days twice a day.After 42 days, mechanical plaque control was interrupted for 5 days. The clinical parameters of gingivitis; Plaque index (PI), gingival index (GI), probing bleeding (BOP), probing depth (PPD) were recorded at baseline, day 42 (beginning of experimental gingivitis) and day 47 (the end of experimental gingivitis). At the same time points, gingival crevicular fluid had been collected for analysis of matrix metalloproteinase - 8 (MMP-8).

DETAILED DESCRIPTION:
The most used and studied probiotics in the periodontal literature are lactobacillus and bifidobacterium. The current study aims to observe the effects of daily ayran consumption containing a probiotic combination of Lactobacillus acidophilus and Bifidobacterium bifidum on plaque development and gingival inflammation in an experimental gingivitis model of healthy individuals. The null hypothesis of this study using of probiotics has no additional benefit for periodontal health.

This study evaluates the effects of daily consumption of ayran containing a probiotic combination of Lactobacillus Acidophilus and Bifidobacterium Bifidum on plaque development and gingival status in healthy individuals with experimental gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Systemic healthy
* Subjects with gingivitis defined as a BOP sites ≥ 10% and PD ≤ 3 mm
* No radiographic bone loss
* Non-smoking participants

Exclusion Criteria:

* History of using antibiotics or anti-inflammatory drugs or probiotic preparations or food supplements in the last 6 months,
* Undergoing orthodontic treatment,
* Active carious lesions
* Mouth breathing
* History of allergy for milk or fermented milk products.
* Taking medications affecting the gingiva and/or oral mucosa

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Plaque index | Plaque index will be recorded at baseline, at day 42 and 47
  PI was scored from 0 to 5 according to the color change obtained with the Mira-2 solution
Gingival index | Gingival index will be recorded at baseline, at day 42 and 47
  GI is graded by visual assessment and mechanical stimulation of the gingival tissues, scoring the gingival condition according to the criteria
Bleeding on probing | BOP will be recorded at baseline, at day 42 and 47
  The probing bleeding (BOP) index was determined by the presence/absence of bleeding ≈30 seconds after probing

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Haytac, phd, Principal Investigator — Professor Doctor
Locations (1):
- Cukurova University Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared upon request
Supporting Information: Study Protocol
Time Frame: The data is ready and can be shared for two years
Access Criteria: The data will be shared upon request